CLINICAL TRIAL: NCT01840631
Title: A Randomized Controlled Trial To Study The Effects Of Group Versus Individual Dietary Counseling In Pediatric Obesity
Brief Title: A Trial To Study The Effects Of Group Versus Individual Dietary Counseling In Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Lisa Underland, Asst. Professor, Pediatrics, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-214
Record Dates: First submitted 2013-03-08; First posted 2013-04-26 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: Obesity; Nutritional counseling; Physical activity; Food diary
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group nutritional counseling (Active Comparator): In this arm, the Nutritionist will conduct the nutritional counseling with numerous patient families as a group
  Interventions: Behavioral: Nutritional Counseling
- Individual nutritional counseling (Active Comparator): In this arm the nutritionist conducts the nutritional counseling with one patient family at a time
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — Participants enrolled will be randomized into group nutrition counseling or individual nutrition counseling classes, for a total of 6 classes. Classes will meet one time a month. Classes will cover topics including nutrition, exercise, and behavior to promote healthy eating.

SUMMARY:
Aim 1 - The primary aim of the study is to assess whether group counseling is a non-inferior intervention compared to the usual care of individual counseling in the management of childhood obesity. In order to achieve this aim, the investigators will compare the mean change in BMI after 6 months of intervention in the two study arms.

Aim 2 - The secondary aim of the study is to determine if the change in BMI is associated with changes in the dietary composition, physical activity and metabolic profile.

DETAILED DESCRIPTION:
This is a non-inferiority study to determine the sample size needed for a larger study to explore an intervention strategy focused on nutrition counseling to maximize weight loss and minimize cardiovascular risk factors in obese children and adolescents. This is a prospective parallel arm, randomized trial, to study the impact of nutritional counseling in an individual vs. group setting. There will be a total of four groups. Obese pre-adolescents (ages 9-12) and adolescents (ages 13-17) will be randomized into two interventions: individual nutrition counseling or group nutrition counseling. Subjects will receive the same information in both interventions. All content will be developed prior to starting the intervention. Each group session will have a maximum of 7 children with 1 parent/caregiver per child and a minimum of 5 children with a caregiver. Group sessions will be one time a month for 60 minutes (30 minutes for dietetic session and 30 minutes for discussion/questions) and individual sessions will be one time a month for 30 minutes. There will be 6 sessions for each group.

All groups will receive standard of care for physical fitness counseling which includes recommending 1 hour of physical activity a day and limiting screen time to less than 2 hours a day. All groups will be evaluated for depression and appropriately referred if found to be depressed. Behavioral strategies, like mindful eating, will be included in the nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 9-17 years of age with a BMI percentile for age of ≥95
* Subjects must be able to attend monthly sessions with a parent and/or guardian.

Exclusion Criteria:

* Subjects with diabetes at baseline, mental or psychological disease that would interfere with understanding, disease or medication causing obesity or weight loss, and participants in an alternative weight management program will not be included in the study.
* Subjects with impaired glucose tolerance will not be excluded from participation.
* Non-English speaking subjects will not be excluded.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change I Mean Body Mass Index | Baseline, month 6
  The primary aim of the study is to assess whether group counseling is a non-inferior intervention compared to the usual care of individual counseling in the management of childhood obesity. In order to achieve this aim, investigators will compare the mean change in BMI after 6 months of intervention in the two study arms. As per previous studies, it is expected the group intervention arm to achieve a mean BMI reduction of 0.8 +/- 1.4 greater than the control arm. The study also posits that a difference in mean BMI change as low as 0.1 would be clinically equivalent.

SECONDARY OUTCOMES:
Change in BMI with diet | Baseline, month 6
  The secondary aim of the study is to determine if the change in BMI is associated with changes in the dietary composition. All the secondary outcomes will be measured by Pearson correlation coefficients or multi-variable linear regression models as appropriate to calculate this.
Change in BMI with physical activity | Baseline, month 6
  The study will assess if there is a change in BMI with increased physical activity
Change in BMI with metabolic profile | Baseline, month 6
  Study will assess if the change in BMI affects Metabolic profile of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Underland, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine West Campus CRC, The Bronx, New York, United States